CLINICAL TRIAL: NCT03352557
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability, and Efficacy of BIIB092 in Subjects With Mild Cognitive Impairment Due to Alzheimer's Disease or With Mild Alzheimer's Disease
Brief Title: Phase 2 Study of BIIB092 in Participants With Early Alzheimer's Disease
Acronym: TANGO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study (NCT03352557) was terminated based on lack of efficacy following the placebo-controlled period readout.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 251AD201; 2017-002901-37 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer's Disease
Keywords: Mild cognitive impairment; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — gosuranemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low-dose BIIB092 (Experimental): Intravenous (IV) infusion once every 4 weeks OR once every 12 weeks and placebo at the other 4-week dosing visits to maintain the treatment blind.
  Interventions: Drug: BIIB092
- Medium-dose BIIB092 (Experimental): Intravenous (IV) infusion once every 4 weeks.
  Interventions: Drug: BIIB092
- High-dose BIIB092 (Experimental): Intravenous (IV) infusion once every 4 weeks.
  Interventions: Drug: BIIB092
- Placebo (Placebo Comparator): Intravenous (IV) infusion once every 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB092 — Administered as specified in treatment arm.
  Other Names: Formally known as BMS 986168
  Arms: High-dose BIIB092; Low-dose BIIB092; Medium-dose BIIB092
Drug: Placebo — Administered as specified in treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of the placebo-controlled period is to evaluate the safety and tolerability of BIIB092 in participants with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or with mild AD. The secondary objectives of the placebo-controlled period are to evaluate the efficacy of multiple doses of BIIB092 in slowing cognitive and functional impairment in participants with MCI due to AD or with mild AD, and to evaluate the immunogenicity of BIIB092 after multiple doses in participants with MCI due to AD or with mild AD.

The primary objective of the long-term extension period is to evaluate the long-term safety and tolerability of BIIB092 in participants with MCI due to AD or with mild AD.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a gradual and progressive change in memory function over more than 6 months.
* Must meet all of the clinical criteria for mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or mild AD and must have
* Objective evidence of cognitive impairment at Screening
* Clinical Dementia Rating Scale (CDR) global score of 0.5 for MCI due to AD or 0.5 or 1 for mild AD
* Mini-Mental State Examination (MMSE) score of 22 to 30 (inclusive)
* CDR Memory Box score of ≥0.5
* Must consent to apolipoprotein E (ApoE) genotyping
* Must have 1 informant/study partner
* Must have amyloid beta positivity confirmed at Screening

Key Exclusion Criteria:

* Any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns
* Clinically significant, unstable psychiatric illness
* Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* History of unstable angina, myocardial infarction, chronic heart failure or clinically significant conduction abnormalities within 1 year prior to Screening Visit 1
* Indication of impaired renal or liver function
* Alcohol or substance abuse in past 1 year
* Clinically significant systemic illness or serious infection within 30 days prior to or during the screening period
* Use of allowed medications for chronic conditions at doses that have not been stable for at least 4 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1, or use of AD medications at doses that have not been stable for at least 8 weeks prior to Screening Visit 1 and during the screening period up to Study Day 1.
* Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participants at higher risk for adverse events (AEs), or impair the participant's ability to perform cognitive testing or complete study procedures.
* Contraindications to study procedures

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (101):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Xenoscience Inc, Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Dignity Health, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - The Research Center of Southern California, Carlsbad, California
  - Positron Research International, Fremont, California
  - Neuropain Medical Center, Fresno, California
  - V Royter, MD, APMC, Hanford, California
  - Irvine Center for Clinical Research, Inc., Irvine, California
  - Research Center for Clinical Studies West, Lancaster, California
  - Mary S. Easton Center for Alzheimer's Disease Research, UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Pacific Research Network, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Invicro, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Brain Matters Research, Stuart, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Emory University Cognitive Neurology Clinic & ADRC, Atlanta, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Tufts, Boston, Massachusetts
  - Brigham and Women's Hospital Department of Neurology, Boston, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks, M.D., P.C., Plymouth, Massachusetts
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Enhancement Center of NJ, Toms River, New Jersey
  - New York University Medical Center PRIME, New York, New York
  - AD-CARE, University of Rochester, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Neurology Clinic, PC, Cordova, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The Memory Clinic, Inc., Bennington, Vermont
  - Cognition Health, Fairfax, Virginia
- Australia (5):
  - Box Hill Hospital, Box Hill, Victoria
  - Caulfield Hospital, Caulfield, Victoria
  - Austin Hospital, Heidelberg West, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- France (9):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hôpital La Grave, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Nantes - Hopital Nord Laënnec, Nantes, Loire Atlantique
  - Hôpital Lariboisière, Paris, Paris
  - Hôpital des Chapennes, Villeurbanne, Rhone
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (8):
  - Studienzentrum fur Neurologie und Psychiatrie, Böblingen, Baden-Wurttemberg
  - ISPG - Institut fuer Studien zur Psychischen Gesundheit, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Institut fuer Schlaganfall- und Demenzforschung (ISD), Munich, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - Charite - Campus Berlin Buch, Experimental and Clinical Research Center (ECRC), Berlin
- Italy (5):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo, Palermo
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - ULSS 6 Vicenza, Vicenza
- Japan (6):
  - Research Site, Obu-shi, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Suita-shi, Osaka
- Poland (5):
  - PALLMED Sp. z o.o., Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Centrum Medyczne Senior, Sopot
  - Centrum Medyczne NeuroProtect, Warsaw
  - Mazowiecki Szpital Wojewódzki w Warszawie Sp z oo, Warsaw
- Spain (8):
  - CAE Oroitu, Getxo, Vizcaya
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Fundacio ACE, Barcelona
  - Hospital de Santa Maria, Lleida
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Skånes Universitetssjukhus, Malmo
  - Sahlgrenska Universitetssjukhuset, Mölndal Sjukhus, Mölndal
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Shulman M, Kong J, O'Gorman J, Ratti E, Rajagovindan R, Viollet L, Huang E, Sharma S, Racine AM, Czerkowicz J, Graham D, Li Y, Hering H, Haeberlein SB. TANGO: a placebo-controlled randomized phase 2 study of efficacy and safety of the anti-tau monoclonal antibody gosuranemab in early Alzheimer's disease. Nat Aging. 2023 Dec;3(12):1591-1601. doi: 10.1038/s43587-023-00523-w. Epub 2023 Nov 27. PMID 38012285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at approximately 100 investigational sites from 03 May 2018 to 30 August 2021.
Pre-assignment Details: A total of 654 participants with Alzheimer's Disease (AD) were enrolled and randomized to receive placebo or BIIB092 125/375/600/2000 milligrams(mg) in Placebo-Controlled (PC) period. Following PC period, 521 participants entered and 516 were dosed in Long-term Extension (LTE) period, and no participants completed the study due to early termination of the study. WBP/G=Withdrawal by Parent/Guardian
Groups:
- PC Period: Placebo: Participants received BIIB092-matching placebo, intravenous (IV) infusion, on Day 1 and then once every 4 weeks for 76 weeks during the PC period.
- PC Period: BIIB092 125 mg/4 Week: Participants received BIIB092, 125 mg, IV infusion, on Day 1 and then once every 4 weeks for 76 weeks during the PC period.
- PC Period: BIIB092 375 mg/12 Week: Participants received BIIB092, 375 mg, IV infusion, on Day 1 and then once every 12 weeks for 76 weeks during the PC period.
- PC Period: BIIB092 600 mg/4 Week: Participants received BIIB092, 600 mg, IV infusion, on Day 1 and then once every 4 weeks for 76 weeks during the PC period.
- PC Period: BIIB092 2000 mg/4 Week: Participants received BIIB092, 2000 mg, IV infusion, on Day 1 and then once every 4 weeks for 76 weeks during the PC period.
- LTE Period: BIIB092 125 mg/4 Week: Participants who received BIIB092, 125 mg, IV infusion during the PC period, continued to receive BIIB092, 125 mg, IV infusion once every 4 weeks from Week 80 to Week 155 during the LTE period.
- LTE Period: BIIB092 375 mg/12 Week: Participants who received BIIB092, 375 mg, IV infusion during the PC period, continued to receive BIIB092, 375 mg, IV infusion once every 12 weeks from Week 80 to Week 155 during the LTE period.
- LTE Period: BIIB092 600 mg/4 Week: Participants who received BIIB092, 600 mg, IV infusion during the PC period, continued to receive BIIB092, 600 mg, IV infusion once every 4 weeks from Week 80 to Week 155 during the LTE period.
- LTE Period: BIIB092 2000 mg/4 Week - Early Start: Participants who received BIIB092, 2000 mg, IV infusion during the PC period, continued to receive BIIB092, 2000 mg, IV infusion once every 4 weeks from Week 80 to Week 155 during the LTE period.
- LTE Period: BIIB092 2000 mg/4 Week - Late Start: Participants who received BIIB092-matching placebo, IV infusion during the PC period, received BIIB092, 2000 mg, IV infusion once every 4 weeks from Week 80 to Week 155 during the LTE period.
Period: PC Period: Day 1 to Week 78
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week | LTE Period: BIIB092 125 mg/4 Week | LTE Period: BIIB092 375 mg/12 Week | LTE Period: BIIB092 600 mg/4 Week | LTE Period: BIIB092 2000 mg/4 Week - Early Start | LTE Period: BIIB092 2000 mg/4 Week - Late Start
Started | 214 | 58 | 58 | 106 | 218 | 0 | 0 | 0 | 0 | 0
Safety Analysis Set (Safety Analysis Set = Dosed Participants) | 214 | 58 | 58 | 106 | 214 | 0 | 0 | 0 | 0 | 0
Full Analysis Set (FAS) | 214 | 58 | 58 | 106 | 214 | 0 | 0 | 0 | 0 | 0
Antidrug Antibody (ADA) Evaluable Set | 211 | 57 | 57 | 105 | 212 | 0 | 0 | 0 | 0 | 0
Completed | 172 | 48 | 50 | 91 | 175 | 0 | 0 | 0 | 0 | 0
Not Completed | 42 | 10 | 8 | 15 | 43 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance with Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized by Mistake | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant-Study Visit Burden/Scheduling Conflicts | 7 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant-Concern About Study Procedures/Perceived Risks | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant-Relocation (Moving or Has Moved) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant-Desire for Change in Treatment (Unrelated to Safety) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant-Other | 6 | 2 | 2 | 5 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — WBP/G-Study Visit Burden/Scheduling Conflicts | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — WBP/G-Concern About Study Procedures/Perceived Risks | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — WBP/G-Desire for Change in Treatment (Unrelated to Safety) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — WBP/G-Unable to Continue to Enable Participation due to Illness/Hospitalization/Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — WBP/G-Other | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision-Unrelated to Safety | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not Dosed | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Period: LTE Period: Week 80 to Week 173
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week | LTE Period: BIIB092 125 mg/4 Week | LTE Period: BIIB092 375 mg/12 Week | LTE Period: BIIB092 600 mg/4 Week | LTE Period: BIIB092 2000 mg/4 Week - Early Start | LTE Period: BIIB092 2000 mg/4 Week - Late Start
Started | 0 | 0 | 0 | 0 | 0 | 46 (2 PC completers did not enter LTE.) | 49 (1 PC completer did not enter LTE.) | 90 (1 PC completer did not enter LTE.) | 169 (6 PC completers did not enter LTE.) | 167 (5 PC completers did not enter LTE.)
Safety Analysis Set (Safety Analysis Set = Dosed Participants) | 0 | 0 | 0 | 0 | 0 | 45 | 49 | 89 | 168 | 165
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 46 | 49 | 90 | 169 | 167
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 38 | 49 | 75 | 151 | 154
Not completed — Withdrawal by Participant-Study Visit Burden/Scheduling Conflicts | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 3 | 3
Not completed — Withdrawal by Participant-Relocation (Moving or Has Moved) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Participant-Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
Not completed — WBP/G-Study Visit Burden/Scheduling Conflicts | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — WBP/G-Concern About Study Procedures/Perceived Risks | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — WBP/G-Relocation (Moving or Has Moved) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — WBP/G-Unable to Continue to Enable Participation due to Illness/Hospitalization/Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — WBP/G-Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants included enrolled participants who received a randomization treatment assignment from the Interactive Response Technology (BIIB092 or placebo).
Groups:
- PC Period: Placebo: Participants received BIIB092-matching placebo, IV infusion, on Day 1 and then once every 4 weeks for 76 weeks during the PC period.
- Total: Total of all reporting groups
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week | Total
Number analyzed (Participants) | 214 | 58 | 58 | 106 | 218 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (6.63) | 70.4 (6.80) | 70.3 (6.79) | 69.7 (6.66) | 69.4 (7.11) | 69.7 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 28 | 26 | 55 | 114 | 329
  Male | 108 | 30 | 32 | 51 | 104 | 325
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 1 | 9 | 17
  Not Hispanic or Latino | 208 | 53 | 55 | 103 | 208 | 627
  Unknown or Not Reported | 3 | 3 | 1 | 2 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 5 | 3 | 2 | 6 | 7 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 1 | 1 | 7
  White | 201 | 53 | 53 | 98 | 206 | 611
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 2 | 1 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: PC Period: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in participant or clinical investigation participant administered pharmaceutical product and that does not necessarily have causal relationship with this treatment. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of medicinal (investigational) product, whether or not related to medicinal (investigational) product. SAE is any untoward medical occurrence that at any dose, results in death; in view of investigator places participant at immediate risk of death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in congenital anomaly/birth defect; is medically important event. Participants who completed treatment period in PC period and did not enter LTE period were to be assessed at Week 90 (14 weeks after end of treatment) as safety follow-up.
Time Frame: Day 1 to Week 78 (participants who entered LTE period); Day 1 up to Week 90 (participants who did not LTE period)
Population: The safety analysis set included all randomized participants who received at least one dose of study treatment (BIIB092 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week
Number analyzed (Participants) | 214 | 58 | 58 | 106 | 214
percentage of participants
  AEs | 84.6 | 86.2 | 82.8 | 88.7 | 88.3
  SAEs | 12.1 | 10.3 | 10.3 | 12.3 | 11.7

2. Primary Outcome: LTE Period: Percentage of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose, results in death; in the view of the investigator places the participant at immediate risk of death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is a medically important event.
Time Frame: From Week 80 to Week 173
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LTE Period: BIIB092 125 mg/4 Week | LTE Period: BIIB092 375 mg/12 Week | LTE Period: BIIB092 600 mg/4 Week | LTE Period: BIIB092 2000 mg/4 Week - Early Start | LTE Period: BIIB092 2000 mg/4 Week - Late Start
Number analyzed (Participants) | 45 | 49 | 89 | 168 | 165
percentage of participants
  AEs | 68.9 | 55.1 | 58.4 | 61.3 | 60.0
  SAEs | 11.1 | 2.0 | 10.1 | 6.0 | 7.9

3. Secondary Outcome: PC Period: Change From Baseline Over Time at Week 78 on the Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score
Description: The CDR-SB is a validated clinical assessment of global function in participants with AD. The CDR is comprised of 6 domains: Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care. CDR-SB is the sum of the scores for these 6 domains. Impairment is scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or "box scores", can be added together to give the CDR-SB score which ranges from 0 (none) to 18 (severe impairment).
Time Frame: Baseline, Week 78
Population: FAS included all randomized participants who received study treatment (BIIB092 or placebo). As pre-specified in study protocol, 125 mg and 375 mg groups were pooled as 'Low dose' group for efficacy analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PC Period: BIIB092 Low Dose: Participants received BIIB092, 125 mg, IV infusion, on Day 1 and then once every 4 weeks or BIIB092, 375 mg, IV infusion, on Day 1 and then once every 12 weeks for 76 weeks during the PC period.
Arm/Group | PC Period: Placebo | PC Period: BIIB092 Low Dose | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week
Number analyzed (Participants) | 214 | 116 | 106 | 214
score on a scale
  Baseline | 3.07 (1.467) | 2.92 (1.620) | 3.24 (1.557) | 3.04 (1.378)
  Change at Week 78: number analyzed (Participants) | 170 | 98 | 91 | 174
  Change at Week 78 | 1.71 (2.376) | 2.10 (2.375) | 2.23 (2.987) | 1.76 (2.038)

4. Secondary Outcome: PC Period: Percentage of Participants With Anti-BIIB092 Antibodies in Serum
Time Frame: Baseline up to Week 76
Population: The ADA evaluable set is defined as participants in the FAS who have an evaluable postbaseline ADA sample.
Measure: Number; unit: percentage of participants
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week
Number analyzed (Participants) | 211 | 57 | 57 | 105 | 212
percentage of participants | 1.9 | 0 | 0 | 1.0 | 0

ADVERSE EVENTS:
Time Frame: From first dose through 14 weeks after last dose of study drug (Up to approximately 173 weeks)
Description: The safety analysis set included all randomized participants who received at least one dose of study treatment (BIIB092 or placebo). The all-cause mortality data and adverse events are reported for 'safety analysis set'.
Arm/Group | PC Period: Placebo | PC Period: BIIB092 125 mg/4 Week | PC Period: BIIB092 375 mg/12 Week | PC Period: BIIB092 600 mg/4 Week | PC Period: BIIB092 2000 mg/4 Week | LTE Period: BIIB092 125 mg/4 Week | LTE Period: BIIB092 375 mg/12 Week | LTE Period: BIIB092 600 mg/4 Week | LTE Period: BIIB092 2000 mg/4 Week - Early Start | LTE Period: BIIB092 2000 mg/4 Week - Late Start
All-Cause Mortality (participants affected / at risk) | 1/214 | 1/58 | 0/58 | 0/106 | 1/214 | 2/45 | 0/49 | 1/89 | 1/168 | 1/165
Serious Adverse Events (participants affected / at risk) | 26/214 | 6/58 | 6/58 | 13/106 | 25/214 | 5/45 | 1/49 | 9/89 | 10/168 | 13/165
Other Adverse Events (participants affected / at risk) | 121/214 | 39/58 | 38/58 | 68/106 | 139/214 | 10/45 | 11/49 | 19/89 | 28/168 | 29/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PC Period: Placebo (N=214) | PC Period: BIIB092 125 mg/4 Week (N=58) | PC Period: BIIB092 375 mg/12 Week (N=58) | PC Period: BIIB092 600 mg/4 Week (N=106) | PC Period: BIIB092 2000 mg/4 Week (N=214) | LTE Period: BIIB092 125 mg/4 Week (N=45) | LTE Period: BIIB092 375 mg/12 Week (N=49) | LTE Period: BIIB092 600 mg/4 Week (N=89) | LTE Period: BIIB092 2000 mg/4 Week - Early Start (N=168) | LTE Period: BIIB092 2000 mg/4 Week - Late Start (N=165)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Idiopathic orbital inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PC Period: Placebo (N=214) | PC Period: BIIB092 125 mg/4 Week (N=58) | PC Period: BIIB092 375 mg/12 Week (N=58) | PC Period: BIIB092 600 mg/4 Week (N=106) | PC Period: BIIB092 2000 mg/4 Week (N=214) | LTE Period: BIIB092 125 mg/4 Week (N=45) | LTE Period: BIIB092 375 mg/12 Week (N=49) | LTE Period: BIIB092 600 mg/4 Week (N=89) | LTE Period: BIIB092 2000 mg/4 Week - Early Start (N=168) | LTE Period: BIIB092 2000 mg/4 Week - Late Start (N=165)
Constipation (Gastrointestinal disorders) | 8 | 5 | 1 | 2 | 6 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 11 | 3 | 6 | 11 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 4 | 2 | 6 | 11 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 7 | 1 | 4 | 8 | 12 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 22 | 4 | 6 | 9 | 24 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 15 | 5 | 3 | 6 | 15 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 13 | 5 | 3 | 8 | 20 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 9 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 23 | 6 | 11 | 19 | 30 | 5 | 7 | 6 | 14 | 15
Contusion (Injury, poisoning and procedural complications) | 6 | 0 | 1 | 8 | 5 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 4 | 2 | 3 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 6 | 7 | 9 | 19 | 0 | 3 | 4 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 5 | 3 | 9 | 13 | 3 | 0 | 2 | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 13 | 5 | 2 | 9 | 11 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 20 | 1 | 6 | 11 | 22 | 1 | 3 | 4 | 3 | 6
Anxiety (Psychiatric disorders) | 11 | 4 | 2 | 3 | 15 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 5 | 4 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 13 | 4 | 2 | 4 | 11 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 2 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 7 | 16 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 14 | 5 | 3 | 6 | 13 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated based on lack of efficacy following the placebo-controlled period readout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (3):
  • Study Protocol (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT03352557/Prot_000.pdf
  • Statistical Analysis Plan: Placebo-Controlled Period (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT03352557/SAP_002.pdf
  • Statistical Analysis Plan: Long-Term Extension Period (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03352557/SAP_003.pdf